CLINICAL TRIAL: NCT04879433
Title: Prospective Open Label Evaluation of Cenobamate Adjunctive Treatment of Adults With Refractory Focal Epilepsy: a "Real-world Experience" Study.
Brief Title: Prospective Open-label Evaluation of Cenobamate Adjunctive Treatment of Adults With Refractory Focal Epilepsy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mid-Atlantic Epilepsy and Sleep Center, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: maesc010
Record Dates: First submitted 2020-12-31; First posted 2021-05-10 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Focal Epilepsy
Keywords: cenobamate,; adjunctive therapy; focal epilepsy
MeSH Terms: conditions — Epilepsies, Partial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the efficacy, safety and tolerability of cenobamate as adjunctive treatment of refractory focal epilepsy

DETAILED DESCRIPTION:
The purpose of the study is to evaluate efficacy and safety of adjunctive cenobamate treatment of adults with drug-resistant focal epilepsy in "real world" clinical setting, providing "real world experience" to help guide future cenobamate treatment. This will be an open label study comparing seizure frequency during 52 weeks of baseline observation period with seizure frequency during 52 weeks of adjunctive cenobamate maintanance treatment. ~100 adults aged 18-70 with severe refractory focal epilepsy with focal seizures that have failed to respond to ≥ 4 antiseizure drugs (ASDs) +/- respective surgery +/- vagal nerve stimulator (VNS), responsive nerve stimulator (RNS) or deep brain stimulator (DBS) treatment with epilepsy duration of ≥ 2 years and followed by the Investigator and/or his epileptologist colleagues at the Investigator's institution for ≥ 1 year will be enrolled. Patients will be on ASDs deemed by the Investigator to have achieved the best seizure control to-date. No more than 5 ASDs will be used. VNS, RNS and DBS will be allowed and not counted as an ASD. However, patients on VNS, RNS or DBS will have to have had the device placed ≥ 6 months before study initiation and have had stable stimulator settings for ≥ 3 months. Baseline will include 52 weeks of prospectively kept, well documented seizure diaries that have been regularly, prospectively reviewed by the treating epileptologist during 52 weeks prior to study initiation. Retrospective review of these diaries will be allowed and count as baseline. As an alternative to seizure diaries, well-documented seizure frequency obtained during regular clinical visits, reviewed by the treating epileptologist and documented in the patient's chart during regular clinical visits during the 52 weeks' baseline period will be allowed in lieu of seizure diaries. ASDs will be held stable during the last month of baseline observation period. Following a baseline of 52 weeks patients will be started on cenobamate, administered orally in qhs, qd or b.i.d. schedule. Both starting dose and titration schedule up to initial target dose of 100-250 mg will follow FDA approved guidelines.

Cenobamate target dose will range from 100-400 mg/day. Within this range, the target dose will be individualized and will be the dose when seizure freedom, intolerable TEAEs or 400 mg/day is reached, whichever occurs first Maintenance period will start when seizure freedom, 250 mg/day dose or maximum tolerated dose of ≥ 100 mg/day is reached, whichever comes first. Maintenance treatment will last for 52 weeks. Total treatment period may vary between subjects depending on titration and final dose, but maintenance treatment period will be 52 weeks for all subjects. During both titration and cenobamate treatment, reduction of the dose of concomitant other ASDs will be allowed as clinically indicated; increase in the dose of concomitant ASDs will not be allowed, nor will initiation of any new antiseizure therapy other than cenobamate. Initiation of new antiseizure treatment or clinically indicated need for increase of ASD other than cenobamate will end of the active part of the study, although patients will be followed to the end of the 52 week maintenance treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70
2. Focal epilepsy uncontrolled in spite of past or present treatment with four or more anti-seizure drugs (ASDs), with focal aware motor seizures, focal unaware seizures and focal to bilateral tonic clonic seizures.
3. Stable ASD doses for at least 30 days
4. Epilepsy duration for ≥ 2 years
5. Past/current treatment with ≥ 4 ASDs. VNS, RNS and DBS treatment will be allowed and will not count as an ASD. VNS, RNS and DBS setting must be stable for 3 months prior to enrollment.
6. Seizure frequency of ≥1/month for ≥ 10/12 months before treatment initiation

Exclusion Criteria:

1. Primary generalized epilepsy
2. Focal aware non-motor seizures without bilateral tonic-clonic seizures
3. Non-epileptic seizures
4. Progressive neurological disease including neoplasm, CNS degenerative disorders including Alzheimer's disease
5. Any systemic illness or unstable medical condition that might pose additional risk, including renal or liver disease, clinically uncontrolled cardiac disease other unstable metabolic or endocrine disturbances, and active systemic cancer
6. Change in the dose of any ASD within 30 days prior to enrollment
7. Active drug or alcohol dependence or any other factors that, in the opinion of the site investigators would interfere with adherence to study requirements
8. Pregnancy
9. Use of any CNS-active investigational drugs within 1 month of enrollment
10. Resective epilepsy surgery less than 6 months before study initiation
11. Vagal nerve stimulator VNS, RNS or DBS implantation less than 6 months before study initiation
12. Adjustment of VNS, RNS or DBS settings less than 3 months before study initiation
13. Inability or unwillingness of subject or legal guardian/representative to give written informed consent.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Male and female adults aged 18-70 with uncontrolled focal epilepsy
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-06-25 (Actual); Primary Completion 2023-06-25 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
The seizure frequency per 28 days. | seizure count per 28 days, baseline 52 weeks, maintanance period 52 weeks
  comparing seizure frequency per 28 day periods during maintanance treatment vs. baseline
seizure freedom rate | 52 weeks of adjunctive cenobamate maintanance treatment
  rate of seizure-free patients
>75% seizure frequency reduction | seizure count per 28 days, baseline 52 weeks, maintanance period 52 weeks
  rate of patients with >75% seizure frequency reduction, comparing seizure frequency per 28 day periods during maintanance treatment vs. baseline
treatment emergent adverse events rate | 52 weeks of baseline period; whole treatment period
  rate of treatment emergent adverse events
treatment discontinuation rate | 52 weeks of baseline period; whole treatment period
  rate of cenobamate treatment discontinuation

SECONDARY OUTCOMES:
median seizure frequency reduction | 52 weeks of baseline period; 52 weeks of adjunctive cenobamate maintanance treatment
  median seizure frequency reduction evaluation in maintenance period
median seizure frequency reduction | 52 weeks of baseline period; the whole treatment period
  median seizure frequency reduction evaluation in treatment period
seizure severity | 52 weeks of baseline period; 52 weeks of adjunctive cenobamate maintanance treatment
  evaluate a seizure severity composite score
quality of life change | 52 weeks of baseline period; the whole treatment period
  quality of life questionnaire (QOLIE-31-P) scores
seizure-related injuries | 52 weeks of baseline period; the whole treatment period
  seizure-related injuries rate
driving status | 52 weeks of baseline period; the whole treatment period
  rate of patients with changed driving status

CONTACTS AND LOCATIONS:
Locations (1):
- Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland, United States